CLINICAL TRIAL: NCT00893360
Title: A Phase I Randomized, Dose Escalation Study of the Safety and Efficacy of Intracoronary Delivery of Cardiosphere-Derived Stem Cells in Patients With Ischemic Left Ventricular Dysfunction and a Recent Myocardial Infarction
Brief Title: CArdiosphere-Derived aUtologous Stem CElls to Reverse ventricUlar dySfunction
Acronym: CADUCEUS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Johns Hopkins University (Other); The Emmes Company, LLC (Industry)
Responsible Party: Principal Investigator, Eduardo Marban, MD, PhD, Director, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IND 13930; U54HL081028 (NIH)
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2012-02

CONDITIONS: Recent Myocardial Infarction; Ventricular Dysfunction
Keywords: Adult Stem cells; Cardiosphere derived stem cells; Myocardial infarction
MeSH Terms: conditions — Ventricular Dysfunction; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cardiac Stem Cell Treatment - Group 1 (Experimental): Autologous stem cell infusion of 12.5 MIL CDCs via intracoronary infusion.
  Interventions: Biological: Autologous stem cell infusion
- Cardiac Stem Cell Treatment -Group 2 (Experimental): Autologous stem cell infusion of 25 MIL CDCs via intracoronary infusion.
  Interventions: Biological: Autologous stem cell infusion
- Observation (Control Group) (No Intervention): Observation of myocardial recovery after usual medical management.

INTERVENTIONS:
Biological: Autologous stem cell infusion — Subjects will receive 12.5 million of autologous (grown from your own heart muscle specimen) cardiosphere-derived stem cells via intracoronary delivery.
  Arms: Cardiac Stem Cell Treatment - Group 1
Biological: Autologous stem cell infusion — Subjects will receive 25 million of autologous (grown from your own heart muscle specimen) cardiosphere-derived stem cells via intracoronary delivery.
  Arms: Cardiac Stem Cell Treatment -Group 2

SUMMARY:
The purpose of this study is to determine whether giving cardiosphere-derived stem cells (CDCs) to patients with decreased heart function and/or a large amount of damaged muscle after a heart attack is safe. CDCs are cells grown from small biopsy samples taken from the heart. Giving a patient their own CDCs is an investigational procedure that has been approved by the Food and Drug Administration for this study. In addition to determining whether this treatment is safe, the study will also examine whether it can decrease the amount of heart muscle damage and/or improve heart function after a heart attack. The amount of heart muscle damage and the function of the heart directly affects prognosis (the predicted course of the disease), and the development of heart failure and other complications some patients experience after a heart attack.

By way of background, scientists and physicians believed, until just a few years ago, that heart muscle damaged after a heart attack could not be replaced. Recently, however, scientists discovered that new heart muscle can form, or be regenerated, and that this process can be enhanced (or increased) by the administration of large numbers of certain cells isolated from the heart or bone marrow. These cells can be stem cells, or cells derived from stem cells, and they may achieve their benefit by forming new heart muscle cells, becoming heart muscle cells themselves, or releasing substances which increase the ability of already existing stem cells to form new heart muscle. All of the studies conducted so far have been experimental and no cell type is approved for routine clinical care of patients with heart disease. However, studies involving bone marrow stem cells do indicate some small improvement in heart function and one large study demonstrated a decrease in clinical events in the group which received bone marrow cells.

Investigators of this study decided to study CDCs because they come from a person's own body, and therefore have no foreign immune antigens which may be rejected. Since the cells come from the person's heart, they are more likely to form heart tissue. In addition, animal studies indicate no safety problems and that these cells are capable of forming heart muscle and blood vessel cells after heart attacks. The investigators are now studying whether the same is true in humans.

DETAILED DESCRIPTION:
The type of study that is being proposed is called a prospective, randomized, dose escalation study. This means that some of the patients will receive a solution which contains the cells and some of the patients will receive conventional medical treatment. The ratio is 2:1, which means that twice as many patients will receive cells as will receive conventional medical treatment. The first 6 patients in each group will be randomized to receive the study drug at a dose of 12.5 million cells or conventional medical treatment. The remaining 18 patients will be randomized to receive study drug at a dose of 25 million cells or conventional medical treatment. The DSMB will evaluate unblinded AE data (including SAEs) when the first six patients have been enrolled and those receiving cells have been discharged. There are two study sites. Each site will enroll 15 participants. The total number of subjects will be 30, with an approximate 20% attrition rate.

Subjects will be referred to participate in the study by physicians caring for them. The target number of participants is 24 patients who have an open artery to inject the stem cells and whose biopsy tissues have been grown to 12.5 million cells. If for some reason the cells cannot be expanded to 12.5 million or the subject's artery is not open enough to allow proper injection, the subject will be replaced in the study population of 24 patients but continue to be followed. This means that the subject will undergo all tests, procedures (except cell infusion) and follow-up visits that would have otherwise been required for participation in the study.

When a subject is determined to be eligible for the study, the protocol will be reviewed with the subject and informed consent will be obtained by a physician participating in the study prior to any testing or treatment.

This study is being conducted at the Cedars-Sinai Medial Center and The Johns Hopkins Hospital. The total length of a subject's participation in the study will be approximately 14 months, from enrollment to 12 month follow-up visit.

SCREENING PHASE - Participants will undergo a screening evaluation. A physical examination with medical history will be performed which includes medication review as well as alcohol or drug use. A blood specimen will be obtained, approximately three teaspoons, to assess for blood counts, chemistry, HIV, hepatitis and pregnancy test for females of childbearing age. An MRI scan will be performed to determine whether the portion of the heart from which the biopsy would be obtained was damaged from the heart attack. MRI will also detect if any cardiac tumors are present. An electrocardiogram will be performed to assess your heart's electrical activity. Additionally, a computed tomography (CT) scan of the chest, abdomen and pelvis will be performed to detect any existing cancer or tumors. If any of the tests are positive, the subject will not be able to participate in the study.

RANDOMIZATION - After the screening visit is completed, subjects will be randomized to either cell infusion or conventional medical therapy. Randomization is 2:1, meaning that twice as many subjects will be randomized to receive cell infusion as conventional medical therapy. Conventional medical therapy after a heart attack can include beta blockers, aspirin, diuretics, cholesterol lowering agents, anticoagulants, ACE inhibitors or calcium channel blockers and enrollment in a cardiac rehabilitation program. Depending on the degree of heart damage and it's affects on the patient's heart rhythm, the patient may be eligible for pacemaker or implantable cardioverter-defibrillator. The specific medical management is determined by the patient's primary care physician or cardiologist.

BASELINE VISIT- At this visit several tests will be performed to assess the heart's baseline function, i.e., the function before cells are infused. It will be conducted prior to the biopsy. These include completion of a questionnaire about how much activity the subject can perform; blood studies to measure blood count and the function of the liver and kidneys; an electrocardiogram which measures the electrical activity of the heart; an exercise test which will also measure blood pressure, heart rate, electrocardiogram, and the amount of oxygen and carbon dioxide in the exhaled air; a test which measures how much distance the subject can walk in six minutes; a test of lung function; a recording of the heart's rhythm over 48 hours; and an MRI to provide information about the baseline function and recovery of the heart since the myocardial infarction.

BIOPSY PHASE - For subjects randomized to receive stem cells, a biopsy of the heart will be performed in the catheterization laboratory. In this test, a small amount of tissue is removed from the internal lining of the heart. A long, flexible tube (catheter), called a bioptome, is inserted into a vein and threaded into the right side of the heart. Most often the catheter is threaded through the jugular vein of the neck under local anesthesia. The tip of the catheter is fitted with tiny jaws that allow the doctor to take very small snips of muscle for microscopic examination. The doctor will take 5-10 small pieces of heart tissue from the right side of the wall that separates the right side of the heart from the left side of the heart. This will be used to grow the cells over a four week period. Blood pressure and vital signs status will be monitored during and for several hours following the procedure. An electrocardiogram; blood (approximately 15 cc or 3 teaspoons) will be obtained to measure your blood count, kidney and liver function; and urine specimen for urinalysis will be collected. An echocardiogram will be performed before the patient leaves the hospital to determine whether the instrument obtaining the biopsy caused a hole in the wall from which the biopsy was obtained.

INTRACORONARY INFUSION PHASE - During this phase, subjects randomized to receive cells will be brought to the cardiac catheterization laboratory to undergo a cardiac catheterization procedure similar to the angioplasty performed to treat the heart attack. However, rather than having an angioplasty, the cells will be injected into the coronary artery whose blockage was responsible for the heart attack. The cells will be infused through a balloon catheter inflated at the previously implanted stent. There will be no new stent implanted unless it is felt clinically necessary. Following the procedure, the subject will remain in the hospital for 24 hours at which time laboratory studies, including cardiac enzymes to rule out cardiac injury, or a heart attack, as well as ECG monitoring will be performed. The subject will be released from the hospital and asked to wear an ECG recording device for 48 hours.

FOLLOW UP VISITS - For all subjects enrolled in the study, there will be six follow-up visits. This is necessary to obtain and compare information from both sets of study participants. Additionally, it is necessary to obtain the information to determine the safety of the cell infusion and whether it has decreased the amount of the heart which is damaged, improved the blood flow and function of the heart and the portion of the heart which received the cells.

A history and physical will be performed at all of the 6 visits, asking the subject about any side effects they may have had and what other medicines they are taking. Additionally, study staff will perform an electrocardiogram, obtain blood and urine studies measuring blood counts and kidney and liver function, and obtain a 48-hour recording of the subject's electrocardiogram. During the six and twelve month visits, a cardiac MRI scan will also be performed to measure the amount of the heart which is damaged and the blood flow and function of the heart and to assess the portion of the heart which received the cells. It will also determine whether any tumors have formed in the heart. At these visits, there will also be a test of lung function, a six-minute walk test, and questions about how much activity the subject can perform. Additionally, there will be an exercise test which will include measuring heart rate, blood pressure, electrocardiogram, and amount of oxygen and carbon dioxide in exhaled air. Patients who receive an implantable cardio-defibrillator during the study will have a cardiac CT instead of MRI.

The patient will be followed in the study for a total of 12 months from the baseline visit and any unexpected effects of the study will be reported to the hospital's institutional review board, the study data safety monitoring board and the FDA, as appropriate, depending on the severity of the adverse event.

ELIGIBILITY:
Inclusion Criteria

* Myocardial infarction due to coronary artery atherosclerotic disease. Myocardial infarction will be defined by a rise in serum troponin I to greater than the 99th percentile of the upper limits of normal with at least one of the following:

  * symptoms of ischemia
  * ECG changes indicative of new ischemia (new ST-T changes or new left bundle branch block)
  * development of pathological Q waves on the ECG
  * imaging evidence of new loss of viable myocardium, OR
  * new regional wall motion abnormality.
* An area of regional dysfunction, i.e., hypokinetic, akinetic, or dyskinetic, as assessed by echocardiography, left ventriculography, or MRI.
* History of successful angioplasty and stent placement, with resultant TIMI grade flow ≥ 2, in the artery supplying the infarcted, dysfunctional territory and through which the cells will be infused.
* Left ventricular ejection fraction of ≥ .25 and ≤ .45 as determined by clinically-indicated assessment of cardiac function (echocardiogram, gated blood pool scan, x-ray contrast ventriculography, CT and/or MRI one day or more following successful reperfusion).
* No further revascularization clinically indicated at the time the patient is assessed for participation in the clinical trial. This will be determined by a cardiologist who is not an investigator in the clinical trial. No further revascularization may be indicated by no arteries with significant stenosis, the location, and extent of any stenosis may not be suitable for angioplasty, the distal vessels may not be suitable for placement of bypass grafts, and/or the patient declines angioplasty or bypass surgery.
* Ability to provide informed consent and follow-up with protocol procedures.
* Age > 18 years.

Exclusion Criteria:

* Non-cardiovascular disease with expected life expectancy of < 3 years.
* Contraindications to MRI, including:

  * prior ICD placement
  * estimated glomerular filtration rate < 50 ml/min
  * known reaction to gadolinium
  * claustrophobia
  * pacemaker
  * ear implant, and cochlear implant.
* History of possible presence of ferromagnetic material including programmable shunt, shrapnel, penile prosthesis, intra-uterine device, bullets, tattoos, artificial limb, blood vessel coil, and tissue expander may require special screening.
* Septal infarction involving the right ventricular endocardium as demonstrated by screening MRI (because its presence might increase the potential risk of septal biopsy and decrease treatment benefit due to decreased viability of injured septal-based stem cells).
* History of cardiac tumor, or cardiac tumor demonstrated on MRI.
* Requirement for chronic immunosuppressive therapy.
* Participation in an on-going protocol studying an experimental drug or device.
* Diagnosis of right ventricular arrhythmogenic dysplasia.
* Patients with occlusion of the infarct-related artery before administration of the study agent.
* Current alcohol abuse.
* Current drug abuse.
* Pregnancy.
* Child-bearing potential without use of effective contraception. Men intending to "father" children are also excluded.
* Human Immunodeficiency virus infection.
* Viral hepatitis.
* Uncontrolled diabetes and/or hemoglobin A1C > 8.5%.
* Abnormal liver function (SGPT > 3 times the upper reference range) and hematology (hematocrit < 25%, WBC < 3000, platelets < 100,000) studies without a reversible, identifiable cause.
* Ventricular tachycardia or fibrillation not associated with an acute ischemic episode.
* New York Heart Association Class 4 congestive heart failure.
* Canadian Cardiovascular Society Angina Class 3 or 4.
* Evidence of tumor on screening chest/abdominal/pelvic (body) CT scan.
* Symptomatic ventricular tachyarrhythmia complicating the index myocardial infarction.
* Individuals who are not fluent in English.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-05; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The primary objective is to demonstrate the safety of autologous cardiosphere-derived stem cells administered by intra-coronary infusion in patients with ischemic left ventricular dysfunction and a recent myocardial infarction. | 6 months

SECONDARY OUTCOMES:
The secondary objective is to demonstrate the efficacy of autologous cardiosphere-derived cells administered by intra-coronary infusion in patients with ischemic left ventricular dysfunction and a recent myocardial infarction. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Marban, MD, PhD, Principal Investigator — The Heart Institute, Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Johns Hopkins Hospital, Baltimore, Maryland

REFERENCES:
- [Result] Makkar RR, Smith RR, Cheng K, Malliaras K, Thomson LE, Berman D, Czer LS, Marban L, Mendizabal A, Johnston PV, Russell SD, Schuleri KH, Lardo AC, Gerstenblith G, Marban E. Intracoronary cardiosphere-derived cells for heart regeneration after myocardial infarction (CADUCEUS): a prospective, randomised phase 1 trial. Lancet. 2012 Mar 10;379(9819):895-904. doi: 10.1016/S0140-6736(12)60195-0. Epub 2012 Feb 14. PMID 22336189
- [Derived] Malliaras K, Makkar RR, Smith RR, Cheng K, Wu E, Bonow RO, Marban L, Mendizabal A, Cingolani E, Johnston PV, Gerstenblith G, Schuleri KH, Lardo AC, Marban E. Intracoronary cardiosphere-derived cells after myocardial infarction: evidence of therapeutic regeneration in the final 1-year results of the CADUCEUS trial (CArdiosphere-Derived aUtologous stem CElls to reverse ventricUlar dySfunction). J Am Coll Cardiol. 2014 Jan 21;63(2):110-22. doi: 10.1016/j.jacc.2013.08.724. Epub 2013 Sep 11. PMID 24036024
- [Derived] Wang S, Li R, Fettermann A, Li Z, Qian Y, Liu Y, Wang X, Zhou A, Mo JQ, Yang L, Jiang P, Taschner A, Rossmanith W, Guan MX. Maternally inherited essential hypertension is associated with the novel 4263A>G mutation in the mitochondrial tRNAIle gene in a large Han Chinese family. Circ Res. 2011 Apr 1;108(7):862-70. doi: 10.1161/CIRCRESAHA.110.231811. PMID 21454794
- [Derived] D'Amario D, Fiorini C, Campbell PM, Goichberg P, Sanada F, Zheng H, Hosoda T, Rota M, Connell JM, Gallegos RP, Welt FG, Givertz MM, Mitchell RN, Leri A, Kajstura J, Pfeffer MA, Anversa P. Functionally competent cardiac stem cells can be isolated from endomyocardial biopsies of patients with advanced cardiomyopathies. Circ Res. 2011 Apr 1;108(7):857-61. doi: 10.1161/CIRCRESAHA.111.241380. Epub 2011 Feb 17. PMID 21330601